CLINICAL TRIAL: NCT04191837
Title: Self-administered Acupressure for Knee Osteoarthritis in Middle- and Older-Aged Adults: A Randomized Controlled Trial
Brief Title: Self-administered Acupressure for Knee Osteoarthritis in Middle- and Older-Aged Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Self-Acup KneeOA
Record Dates: First submitted 2019-09-17; First posted 2019-12-10 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-administered acupressure (Experimental): A training course will be offered to subjects in this group to train them to perform self-acupressure.
  Interventions: Other: Self-administered acupressure treatment group
- Knee health education (Active Comparator): A course regarding knee health will be offered to the subjects in this group.
  Interventions: Other: Knee health education control group

INTERVENTIONS:
Other: Self-administered acupressure treatment group — Subjects in the self-administered acupressure exercise group will receive two training sessions (2 hours each, 1-week apart). The self-administered acupressure treatment protocol was developed based on Chinese medicine meridian theory by previous studies and modified. The acupoints are indicated for knee pain and have been commonly used and tested for feasibility in pilot study. The training will be conducted in a group format with 4-6 subjects per group. Each subject will then receive a handout and an acupressure log. They will be told to perform the self-acupressure twice per day for 12 weeks.The capability of participants for self-administered acupressure will be inspected by the instructor with a competency checklist in each session. And a demonstration video will be sent to the participants via WhatsApp for their reference at home.
  Arms: Self-administered acupressure
Other: Knee health education control group — Subjects in the health education control group will receive knowledge related to knee OA symptom management. The health education will be conducted in a talk format for 2 hours for two sessions. The course content is developed from the course materials from the websites of Elderly Health Service, Department of Health, Hong Kong SAR and reviewed. Subjects in knee health education group will be told to follow the knee health instruction for 12 weeks.
  Arms: Knee health education

SUMMARY:
This is a randomized controlled trial comparing the short-term and medium-term effect of self-administered and knee health education for relieving knee pain in middle-aged and older adults with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the major causes of physical disability commonly influencing people aged above 50 years. Acupressure is proposed for alleviating knee OA symptoms because of the low cost of intervention, accessibility, and safety.

Objectives: 1. To examine the short- and medium-term effectiveness of self-administered acupressure taught by a short training course on relieving knee OA pain in middle-aged and older adults. And to evaluate the subjects' compliance with self-administered acupressure for knee OA.

Hypothesis: self-administered acupressure group would have a greater pain relief compared to the knee health education control in subjects with knee OA at week 4 (short-term) and 12 (medium-term).

Design and subjects: A randomized, parallel-group, control trial. 314 subjects with knee OA will be recruited; 157 per group. All eligible subjects will be randomized to either self-administered acupressure or knee health education control group in 1:1 ratio.

Interventions: Subjects in the self-acupressure group will attend two 2-hour training sessions to learn self-acupressure and will practice self-acupressure twice a day for 12 weeks; subjects in the education control group will receive two 2-hour training sessions to learn the health information related to knee OA. They will be told to follow the knee health instructions for 12 weeks.

Main outcome measures: The primary outcome measure is the numerical rating scale for knee pain. Other measures include Western Ontario and McMaster University Osteoarthritis Index (WOMAC), Short-Form Six-Dimension (SF-6D), Timed Up & Go Test (TUG) and Fast Gait Speed (FGS). Acceptability of two training courses will also be evaluated.

Data Analysis: Differences in the questionnaire scores will be examined using a linear mixed-effects model. Intention-to-treat analyses will be conducted. Effect sizes will be computed by dividing the difference in means by the pooled standard deviation. Incremental costs and incremental effects will be compared between the self-acupressure and knee health education groups and and plotted the results in a cost-effectiveness acceptability curve.

ELIGIBILITY:
Inclusion Criteria:

* ethnic Chinese;
* aged 50 years or above;
* ability to comprehend Chinese;
* fulfilling any 3 of the following criteria: i. morning stiffness ≤ 30 min; ii. crepitus on active joint motion; iii. bone tenderness; iv. bone enlargement; or v. no palpable joint warmth (This classification yielded 84% sensitivity and 89% specificity for OA knee diagnosis);
* having knee pain for at least 3 months;
* Knee pain ≥3 on a Likert pain scale from 1-10;
* having a smartphone (or a family member living together having a smartphone) that is compatible to WhatsApp (it is the investigator's experience in the pilot study that most of every subject had been used to using WhatsApp for social communication);
* willing to provide informed consent

Exclusion Criteria:

* medical diagnoses or conditions that preclude individuals from active participation (e.g. bleeding disorders, alcohol or drug abuse);
* knee pain related to other conditions (cancer, fracture, rheumatoid arthritis, rheumatism) as screened according to the red flags for further investigation or referral in the NICE 2014 Guidelines for Osteoarthritis of the knee;
* score < 22 in Hong Kong Montreal Cognitive Assessment (HK-MoCA) indicating cognitive impairment that may prevent understanding of training instructions;
* body mass index over 30, the obese II criteria for Asians (it will be too difficult for the obese subjects to perform acupressure on the acupoints as physical pressure reaching the muscle is required);
* presence of skin lesions or infections at the treatment sites;
* ever had knee replacement surgery;
* pregnancy or contemplating pregnancy;
* ever received acupressure or steroid injection for knee pain over the past 6 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Pain severity numerical rating scale | Week 4
  a single 11-point numeric scale ranges from 0 (no pain) to 10 (greatest pain imaginable) to indicate the pain severity in recent one week.

SECONDARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | Baseline, Week 4, Week 8, Week 12
  The Western and McMaster Universities Osteoarthritis Index (WOMAC, Likert version 3.1). Its score ranges from 0 to 96.
Short Form 6D (SF-6D) | Baseline, Week 4, Week 8, Week 12
  A preference-based measure of health derived from a selection of SF-36 items for economic evaluation. It is used to measure quality of life.
Timed Up & Go Test (TUG) | Baseline, Week 4, Week 8, Week 12
  The TUG test was developed and modified from a clinical measure of balance, including stand up from armchair, walk for 3 meters, turn around, walk back and sit down. The unit will be expressed in m/s.
Fast Gait Speed (FGS) | Baseline, Week 4, Week 8, Week 12
  To tests the time of crossing a marked 10-meter distance at a speed "as quickly as possible but safe". The unit will be expressed in m/s.
Pain severity numerical rating scale | Week 8, Week 12
  a single 11-point numeric scale ranges from 0 (no pain) to 10 (greatest pain imaginable) to indicate the pain severity in recent one week.

OTHER OUTCOMES:
Self-report frequency of pain medication use | Baseline, Week 4, Week 8, Week 12
  Participants were permitted to continue using routine medications and pain medications, and maintain their usual physician visits throughout the study. The unit will be expressed in no. of day taking pain medication.

CONTACTS AND LOCATIONS:
Overall Officials: Wing-Fai Yeung, Principal Investigator — School of Nursing, the Hong Kong Polytechnic University
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yeung WF, Chen SC, Cheung DST, Wong CK, Chong TC, Ho YS, Suen LKP, Ho LM, Lao L. Self-Administered Acupressure for Probable Knee Osteoarthritis in Middle-Aged and Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245830. doi: 10.1001/jamanetworkopen.2024.5830. PMID 38639940